CLINICAL TRIAL: NCT06118736
Title: GUIDed Growth of the Proximal Femur to Prevent Further Hip MigrAtion in CErebral Palsy Patients
Acronym: GUIDANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Merel Roelen, MD, PhD candidate, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PanamaID 10082
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy; Hip Dislocation
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor tenotomy + Temporary Medial Hemi-epiphysiodesis of the proximal femur (Experimental): Standard care + intervention
  Interventions: Procedure: Temporary Medial Hemi-epiphysiodesis of the proximal femur
- Adductor tenotomy (No Intervention): Standard care

INTERVENTIONS:
Procedure: Temporary Medial Hemi-epiphysiodesis of the proximal femur — Temporary Medial Hemi-epiphysiodesis of the proximal femur
  Arms: Adductor tenotomy + Temporary Medial Hemi-epiphysiodesis of the proximal femur

SUMMARY:
In recent literature, the potential of guided growth of the proximal femur to modify hip growth in patients with cerebral palsy has been shown. Using medial hemi-epiphysiodesis of the proximal femur (TMH-PF) morphology of hips at risk of symptomatic (sub)luxation in cerebral palsy (CP) can be changed, aiming to reduce further hip migration and the need for more invasive surgical treatment modalities. Further research is necessary to assess if the results of TMH-PF in combination with adductor tenotomies are significantly better than the results of the current standard of care; adductor tenotomies alone.

The investigators objective is to determine whether guided growth of the proximal femur decreases the risk of further hip migration and need for further surgery in cerebral palsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Spastic CP
* GMFCS level IV-V
* Aged 2-8 years
* At least one hip with an abduction in flexion ≤ 40 degrees
* Migration percentage of 30-50%
* Head shaft angle > 145

Exclusion Criteria:

* Not fit for surgery
* History of bony hip surgery to the affected hip
* Severe acetabular dysplasia defined as a gothic arch, an incongruent joint or an acetabular index > 30 degrees, consistent with A2 and A3 acetabular deformity according to Robin and Graham in an adequately performed radiographs

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | from enrollment to the end of study (8 years)
  The Primary study outcome is treatment failure, defined as:
  * Need for secondary bony hip surgery to the affected hip or progression to hip migration > 50% at 5-year follow-up . An indication for secondary bony surgery will be defined as;
  * Migration percentage > 50% at a minimum of 1 year after surgery, OR
  * An increased migration > 10% in 1 year during follow-up
  * Increase in Acetabular index to > 30 degrees or an increase of more than 5 degrees during follow-up

SECONDARY OUTCOMES:
Radiographic parameters | from enrollment to the end of study (8 years)
  Standardized conventional radiographs, AP and Lauenstein view (frog leg lateral) Pelvic radiographs will be performed according to the standardized protocol as defined by AACPDM
  * Migration percentage (%), change in migration percentage per treatment arm (on baseline and follow-up)
  * Head Shaft angle (HSA) in degrees
  * Acetabular index
  * Melbourne hip classification
  * Pelvic obliquity
  * Positioning of the hemi epiphysiodesis screw in the intervention group
3-dimensional shape analysis of proximal femur | directly postoperative, at 2-year follow-up and at 5-year follow-up
  CT-scans of the hip will be performed in the intervention group directly postoperative, at 2-year follow-up and 5-year follow-up. On these scans the following measurements will be performed:
  * Positioning of the hemi epiphysiodesis screw
  * 3-dimensional proximal femoral shape analysis regarding (change in) sphericity, congruency and head-neck orientation will be performed in patients at 2-year follow-up and at 5-year follow-up.
  * The direction of migration of the hip and acetabular morphology will be determined according to the method described by Brunner et al.
  * Sphericity of the femoral head will be determined by the Mose technique.
CPChild questionnaire | from enrollment to the end of study (8 years)
  "Caregivers Priorities and Child Health Index of Life with Disabilities"
  The CPCHILD™ is a parent completed questionnaire and was developed to help clinicians to identify areas that are impairing a child's quality of life, determine what is most important to the child and caregiver, and monitor the child's progress in a way that is meaningful to the family.
  Minimum value is 0 and maximum value is 100, the higher the score the better the outcome.
CPG questionnaire | from enrollment to the end of study (8 years)
  CPG = "Checklist Pijn Gedrag" (Dutch for Checklist Pain behaviour) A mean pain score will be calculated.
  A minimum value of 0 with a maximum value of 10. Higher scores mean more pain.
Secondary surgical interventions other than bony procedure | from enrollment to the end of study (8 years)
  Screw revision ▪ The following will be used as indications for screw revision in the intervention group throughout the study period:
  * < 1 thread of the screw remaining in the epiphysis, and
  * HSA > 100 degrees
  Repeated soft tissue release.
  ▪ The following will be used as indications for repeated soft tissue releases (adductor and/or psoas tenotomy) in both the intervention and control group throughout the study period:
  * Abduction < 30 degrees, and
  * No indication for bony surgery

OTHER OUTCOMES:
Baseline measurements | At the time of enrollment
  Other patient related measurements that will be obtained at baseline include
  * Age
  * Weight
  * Height
  * GMFCS classification
  * Change in Migration Percentage in the year prior to the adductor tenotomy
  * Use of tone regulation; Baclofen, Artane, Baclofen pump, Selective Dorsal Rhizotomy (SDR

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Tolk, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (5):
- Netherlands (5):
  - Amsterdam UMC, Amsterdam
  - UMC Groningen, Groningen
  - Maastricht UMC, Maastricht
  - Sint Maartenskliniek, Nijmegen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data that underlie the results from the GUIDANCE study and the study protocol will be shared if requested. Data will be available beginning 12 months and ending 5 years following publication of this paper. Data will be available for researchers who provide a methodologically sound scientific proposal, which has been approved by an ethical committee. Proof of the latter should be provided. Analyses should achieve the aims as reported in the approved proposal. Proposals for data should be directed to the corresponding author.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 12 months and ending 5 years following publication of this paper
Access Criteria: Data will be available for researchers who provide a methodologically sound scientific proposal, which has been approved by an ethical committee. Proof of the latter should be provided. Analyses should achieve the aims as reported in the approved proposal.

REFERENCES:
- [Derived] van Stralen RA, Roelen MCR, Moerman S, Witbreuk MMEH, Witlox MA, Ten Ham A, Eygendaal D, Reijman M, Tolk JJ. GUIDANCE study: guided growth of the proximal femur to prevent further hip migration in patients with cerebral palsy-study protocol for a multicentre randomised controlled trial. BMJ Open. 2024 Dec 11;14(12):e091073. doi: 10.1136/bmjopen-2024-091073. PMID 39663160